CLINICAL TRIAL: NCT06992778
Title: Exploring the Effectiveness and Acceptability of Remote Fine-Tuning of Hearing Aids in Danish Adults: A Non-blinded, Non-inferiority Randomized Controlled Trial With an Embedded Qualitative Study
Brief Title: Effectiveness and Acceptability of Remote Fine-Tuning of Hearing Aids in Danish Adults
Acronym: EARFit
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zealand University Hospital (Other)
Collaborators: Interreg (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SJ-1072
Record Dates: First submitted 2025-03-18; First posted 2025-05-28 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-01

CONDITIONS: Hearing Aid; Telehealth; Hearing Aid Fitting; Effectiveness
Keywords: Remote fine-tuning; Teleaudiology; Randomized controlled trial (RCT); Hearing aids; Denmark

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention Group (IG) (Experimental): Remote Fine-Tuning of Hearing Aids Using Smartphone App
  Interventions: Device: Remote fine-tuning of hearing aids
- Control group (CG) (Active Comparator): Face-to-Face Fine-Tuning of Hearing Aids in Clinic
  Interventions: Device: Face-to-face fine-tuning of hearing aids

INTERVENTIONS:
Device: Remote fine-tuning of hearing aids — Remote Fine-Tuning of Hearing Aids allows patients to adjust their hearing aids remotely, without having to visit a clinic. Using a mobile app on the patient's device, real-time adjustments are made based on their feedback, with immediate changes during the session.
  Unlike traditional face-to-face adjustments, this approach lets patients stay in their own familiar surroundings. This helps create a more accurate listening environment, as the adjustments are made based on the sounds they experience in their everyday life.
  Arms: Intervention Group (IG)
Device: Face-to-face fine-tuning of hearing aids — In the clinic, the standard procedure for fine-tuning hearing aids (HAs) involves a face-to-face consultation with an audiologist, typically lasting 30 minutes.
  Arms: Control group (CG)

SUMMARY:
The aim of this clinical trial is to evaluate the effectiveness and user satisfaction of remote fine-tuning of hearing aids compared to traditional face-to-face adjustments. The main questions aims to answer:

- Are hearing aid outcomes (self-reported and objective) similar when using remote fine-tuning compared to face-to-face adjustments?

Researchers will compare remote fine-tuning (using a smartphone app) to traditional face-to-face fine-tuning sessions in a clinical setting.

Participants will:

* Be randomized to either the remote fine-tuning group (intervention group) or the face-to-face adjustment group (control group).
* Attend five scheduled consultations over a 3-month period, including baseline measurements, hearing aid fittings, and follow-up visits.

Participants in the remote fine-tuning group will:

- Set up and use a hearing aid manufacturer's smartphone app to complete fine-tuning sessions from home.

Participants in the face-to-face group will:

- Visit the clinic for in-person fine-tuning appointments.

Data will be collected through questionnaires (e.g., SSQ-12, IOI-HA, and COSI) and objective measures such as the Speech Intelligibility Index (SII) and speech comprehension in noise (DS-FF). Additional qualitative data will be gathered from interviews with participants in the remote fine-tuning group.

DETAILED DESCRIPTION:
In addition to the randomized controlled trial, a separate qualitative substudy is being conducted to explore user experiences related to the intervention. This component involves independently recruited participants who are not enrolled in the RCT. The qualitative substudy is designed to provide contextual insights into the acceptability, usability, and perceived value of remote fine-tuning of hearing aids from the user perspective. Data are collected through semi-structured interviews and/or observations, and findings will be reported separately to complement the RCT outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with hearing loss who desire HA treatment (+18 of age).
* Danish language skills both written and oral.
* Acquisition of digital proficiency in terms of being familiar with operating a smartphone, including navigating menus, opening and closing apps, and interacting with the touchscreen with capabilities for audio and video calls.
* Access to a smartphone that are compatible with manufacturers' system requirements.
* Access to a stable network connection on the mobile device, with either Wi-Fi or mobile data.

Exclusion Criteria:

* Patients with tinnitus requiring treatment or scoring more than 58 in the 'Tinnitus Handicap Inventory' (THI) grading system.
* Patients with Ménière disease, due to its complications and symptoms as dizziness, balance problems and fluctuating hearing loss, that can affect the HA treatment.
* Patients who will receive in-the-ear (ITE) hearing aids, due to potential limitations in connectivity for remote fine-tuning.
* Patients which are recommended/offered unilateral HA treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-05-27 (Actual); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Self-Reported Hearing Aid Effectiveness | From baseline assessment (2-3 weeks before initial hearing aid fitting) to 12 weeks post-fitting, including all follow-up visits and assessments
  This outcome measures self-reported hearing aid effectiveness using the Speech, Spatial and Qualities of Hearing Scale-12 (SSQ-12)
  Measured at: Baseline (2-3 weeks before hearing aid fitting) and at 12 weeks post-fitting.
  Scoring: SSQ-12 items are rated on a scale of 0-10, with higher scores indicating better hearing perception.
Change from Baseline in Self-Reported Improvement in Hearing | From baseline assessment (2-3 weeks before initial hearing aid fitting) to 12 weeks post-fitting, including all follow-up visits and assessments
  This outcome measures self-reported improvement in hearing using the Client Oriented Scale of Improvement (COSI).
  Measured at: Baseline (2-3 weeks before hearing aid fitting) and at 12 weeks post-fitting.
  Scoring: COSI evaluates improvement in personally relevant listening situations using a five-point scale from "worse" to "much better".
Self-Reported Hearing Aid Satisfaction at 12-Week Follow-Up | At 12-week follow-up, assessing the participant's experience over the past 2 weeks.
  This outcome assesses overall hearing aid satisfaction using the 'International Outcome Inventory for Hearing Aids' (IOI-HA).
  Measured at: 12-week follow-up consultation only.
  Scoring: The IOI-HA consists of 7 items, each designed to assess hearing aid benefit across different domains. Each item is scored on a 1 to 5 scale, where 1 represents the worst outcome and 5 represents the best outcome
Change from Baseline in Speech Intelligibility Index (SII) | Measured at hearing aid fitting and 12 weeks post-fitting.
  This outcome evaluates changes in speech intelligibility using the Aided Speech Intelligibility Index (SII), measured during real-ear-measurement (REM) verification.
  Measured at: Baseline (hearing aid fitting) and at 12-week follow-up.
  Scoring: SII is calculated following ANSI standards (ANSI S3.5-1997), with values ranging from 0 (no speech audibility) to 1.0 (full speech audibility).
Change from Baseline in Discrimination Score in Free Field (DS-FF) | Measured at initial hearing aid fitting and 12 weeks post-fitting.
  This outcome measures changes in speech discrimination ability using the Discrimination Score in Free Field (DS-FF) test under controlled conditions.
  Measured at: Baseline (at initial hearing aid fitting) and at 12-week follow-up.
  Scoring: Speech discrimination performance will be assessed in noise at a speech level of 65 dB SPL. The outcome is expressed as a percentage score (0-100%), where higher percentages indicate better speech discrimination ability. Testing is conducted using DANTALE-1, a validated Danish speech material.

CONTACTS AND LOCATIONS:
Overall Officials: Bjarki Ditlev Djurhuus, MD, PhD, Assoc Prof, Study Chair — Zealand University Hospital
Locations (1):
- Zealand University Hospital, Køge, Denmark

IPD SHARING:
Plan to Share IPD: No